CLINICAL TRIAL: NCT05926583
Title: Phase 3 Study to Evaluate the Safety and Efficacy of AAV5-hRKp.RPGR for the Treatment of Japanese X-linked Retinitis Pigmentosa Associated With Pathogenic Variants in Retinitis Pigmentosa GTPase Regulator (RPGR)
Brief Title: A Study of AAV5-hRKp.RPGR for the Treatment of Japanese Participants With X-linked Retinitis Pigmentosa
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR109143; 74765340RPG3001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: AAV5-hRKp.RPGR Low Dose (Experimental): Participants will receive bilateral subretinal administration of AAV5-hRKp.RPGR low dose, with surgical delivery to the 2 eyes performed within 7 to 21 days apart.
  Interventions: Genetic: AAV5-hRKp.RPGR
- Group 2: AAV5-hRKp.RPGR High Dose (Experimental): Participants will receive bilateral subretinal administration of AAV5 hRKp.RPGR high dose, with surgical delivery to the 2 eyes performed within 7 to 21 days apart.
  Interventions: Genetic: AAV5-hRKp.RPGR

INTERVENTIONS:
Genetic: AAV5-hRKp.RPGR — AAV5-hRKp.RPGR will be administered by subretinal injection using a standardized surgical procedure.
  Arms: Group 1: AAV5-hRKp.RPGR Low Dose
Genetic: AAV5-hRKp.RPGR — AAV5-hRKp.RPGR will be administered by subretinal injection using a standardized surgical procedure.
  Arms: Group 2: AAV5-hRKp.RPGR High Dose

SUMMARY:
The purpose of the study is to assess the safety and tolerability of bilateral subretinal delivery of adeno-associated virus vector with a serotype 5 capsid human rhodopsin kinase promoter. retinitis pigmentosa guanosine triphosphatase regulator (AAV5-hRKp.RPGR).

ELIGIBILITY:
Inclusion Criteria:

* Participants who are Japanese male or female aged 5 years or older
* Participants diagnosed as X-linked retinitis pigmentosa (XLRP) (generalized rod-cone dystrophy) associated with pathogenic or likely pathogenic variants in the retinitis pigmentosa guanosine triphosphatase regulator(RPGR) gene
* Has evidence of preserved retinal function as defined by a mean retinal sensitivity of greater than or equal to (>=) 2 decibel (dB) by Octopus static perimetry and evidence of preserved outer retinal structure (namely the presence of discernible ellipsoid zone) as determined by spectral domain-optical coherence tomography (SD-OCT) in both eyes
* Otherwise, healthy participant on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel or hematology outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator

Exclusion Criteria:

* Has had ocular surgery within 3 months prior to screening or is anticipated to require ocular surgery within 6 months after the AAV5-hRKp.RPGR administration
* Is unable to perform the imaging assessments as required (for example: reliable static perimetry [reliability factor less than or equal to {<=}19], optical coherence tomography [OCT], or fundus autofluorescence [FAF]).
* Any investigational ocular treatment or any other ocular treatment that could confound the interpretation of the efficacy results or affect participant compliance with the visit schedule

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-11-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Event (AEs) | Up to 60 Months
  An AE is any untoward medical occurrence in a clinical study participant administered a investigational or non-investigational medicinal product. An AE does not necessarily have a causal relationship with the treatment.
Number of Participants with Abnormalities in Clinical Laboratory Assessments | Up to 60 Months
  Number of participants with abnormalities in clinical laboratory assessment (hematology and serum chemistry) will be reported.

SECONDARY OUTCOMES:
Change From Baseline in Low Luminance Visual Acuity by Early Treatment Diabetic Retinopathy Study (ETDRS) Chart Letter Score in Monocular Assessment at Week 52 | Baseline - Week 52
  Change from baseline in low luminance visual acuity by ETDRS chart score in monocular assessment at week 52 will be reported.
Change From Baseline in Best Corrected Visual Acuity (BCVA) by Early Treatment Diabetic Retinopathy Study Chart Letter Score in Monocular Assessment at Week 52 | Baseline - Week 52
  Change from baseline in BCVA by ETDRS chart letter score in monocular assessment at week 52 will be reported.
Change From Baseline in Low Luminance Visual Acuity by Early Treatment Diabetic Retinopathy Study Chart Letter Score in Worse-seeing Eye at Week 52 | Baseline - Week 52
  Change from baseline in low luminance visual acuity by ETDRS chart letter score in worse-seeing eye at week 52 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- National Hospital Organization Tokyo Medical Center, Meguro-ku, Japan

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Wang CY, Chen L, Lin TY, Huang SP. Systematic Identification of Candidate Genes for Inherited Retinal Disease Gene Therapy Integrating Worldwide IRD Cohort and Single-Cell Analysis. J Ophthalmol. 2025 Jun 12;2025:7014745. doi: 10.1155/joph/7014745. eCollection 2025. PMID 40547876